CLINICAL TRIAL: NCT05841667
Title: A Clinical Study to Explore the Effect of Carboxylesterase 1 (CES1) Genotype on Pharmacokinetics, Safety, and Efficacy of Remimazolam
Brief Title: Impact of CES1 Genotype on Remimazolam
Status: Recruiting | Type: Observational
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Byung Gun Lim, Professor, Korea University Guro Hospital
Other Study IDs: 2023GR0069
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Adult; Middle Aged; Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CES1 without or without single nucleotide polymorphism (SNP): We will determine the CES1 genotype of participants through a laboratory test. Several different types of SNPs can be identified, and analyses can be further stratified by CES1 SNP type.
  Interventions: Drug: Remimazolam besylate

INTERVENTIONS:
Drug: Remimazolam besylate — This is an observational study, meaning that no interventions are actually administered to the participants. However, blood and urine samples will be collected for research purposes.
  Participants will receive remimazolam besylate for at least 2 hours during anesthesia and surgery. Blood will be drawn to determine the concentration of remimazolam in the blood at the following time points: (1) before remimazolam administration, (2) after remimazolam administration has lasted at least 2 hours without a change in concentration, (3) immediately before discontinuation of remimazolam if there has been a change in concentration since the second blood draw, (4) within 5 minutes of discontinuation, (5) within 15-60 minutes of discontinuation, and (6) 90 minutes after discontinuation. Urine will also be collected after the end of anesthesia to check for metabolites of remimazolam.

SUMMARY:
Remimazolam is primarily metabolized via CES1, and other drugs that are commonly metabolized by CES1 are known to have their pharmacokinetics and clinical effects affected by genetic polymorphisms in CES1.

The goal of this observational study is to investigate the impact of the CES1 genotype on the pharmacokinetics, safety, and efficacy of remimazolam in patients undergoing elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1 or 2
* Age 19-70 years
* Elective surgery

Exclusion Criteria:

* Concomitant regional anesthesia
* Uncontrolled hypertension (systolic blood pressure >180 mmHg)
* Uncontrolled diabetes mellitus (HbA1c >9.0%)
* Aspartate transaminase (AST), Alanine transferase (ALT), Total bilirubin > more than 2 times the normal upper limit
* Estimated glomerular filtration rate <60 ml/min/1.73m2
* Moderate to severe chronic pulmonary obstructive disease or respiratory failure
* Emergency
* Hepatectomy, Liver transplantation
* Cardiopulmonary bypass use
* Craniotomy due to head trauma, unstable intracranial pressure, or brain disease
* Use of benzodiazepine medications (if tolerance is present)
* Anxiety, alcohol/drug dependence, or addiction to tricyclic antidepressants
* Reported hypersensitivity and adverse reactions to benzodiazepines, flumazenil, and other agents used during anesthesia
* Lactose-related genetic disorders
* Myasthenia gravis or myasthenia gravis syndrome
* Newly diagnosed myocardial infarction/clinically significant coronary artery disease, cerebral ischemic attack/stroke within 6 months, or significant untreated coronary artery disease
* Implanted rate-responsive cardiac pacemaker with a bioelectrical impedance sensor.
* Intrinsic brain disorders or other conditions that make it difficult to determine the depth of anesthesia through EEG measurements (e.g., epilepsy)
* History of severe allergies
* Cognitive impairment that prevents comprehension of the instructions and consent form of this study, in case of sedation
* Expected intraoperative blood loss of 1000 ml or more
* Judged by the investigator to be unsuitable for participation in this study due to other reasons

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on adult patients aged 19-70 years, ASA physical status 1-2, undergoing elective surgery in the operating room of Korea University Guro Hospital.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-adjusted steady-state concentration of remimazolam | Immediately before the initiation of remimazolam administration ~ 120 minutes after the cessation of remimazolam
  Determine the dose-adjusted steady-state concentration of remimazolam using Liquid Chromatography-Mass Spectrometry/Mass Spectrometry (LC-MS/MS)
Maintenance dose of remimazolam for maintaining general anesthesia | Immediately before the initiation of remimazolam administration ~ 120 minutes after the cessation of remimazolam
  Hourly maintenance dose of remimazolam for maintaining general anesthesia
Total dose of remimazolam used to induce general anesthesia | Initiation of remimazolam administration ~ 5 minutes after start of remimazolam
  Determine the total dose of remimazolam to achieve loss of consciousness (LOC). Modified Observer's Alertness/Sedation Scale (MOAA/S) <2 indicates LOC. The MOAA/S scale assesses a patient's level of alertness and response to stimulation, and is scored on a 6-point scale (6: awake and alert, 1: deeply asleep and unresponsive to any stimulus).

SECONDARY OUTCOMES:
Time to LOC after remimazolam administration during anesthesia induction | Initiation of remimazolam administration ~ 5 minutes after start of remimazolam
  Determine the time to achieve LOC after remimazolam dosing.
Time to bispectral index(BIS) < 60 after remimazolam administration during anesthesia induction | Initiation of remimazolam administration ~ 10 minutes after start of remimazolam
  Determine the time to achieve BIS <60 after remimazolam dosing
Changes in BIS during induction and maintenance of anesthesia | Initiation of remimazolam administration ~ 30 minutes after cessation of remimazolam
  Measure BIS during anesthesia
Percentage maintained BIS >60 during general anesthesia | Initiation of remimazolam administration ~ Cessation of remimazolam(up to 10 hours after start of remimazolam administration)
  Calculate "Time maintained BIS >60 / Time remimazolam administered"
Changes in BIS during anesthesia induction and maintenance | Initiation of remimazolam administration ~ 30 minutes after cessation of remimazolam
  Assess BIS values during general anesthesia
Postanesthesia care unit (PACU) length of stay | PACU admission ~ PACU discharge (within 3 hours after PACU admission)
  Determine how long participants stay in the PACU before being transferred to a general ward
Emergence delirium | Immediately after extubation ~ 3 hours after PACU admission
  Richmond Agitation Sedation Scale (RASS) ≥1 indicates emergence delirium (RASS score ranges from -5 to +4, with negative numbers indicating varying degrees of sedation or lethargy, and positive numbers indicating varying degrees of agitation or restlessness)
Resedation | Immediately after extubation ~ 3 hours after PACU admission
  Richmond Agitation Sedation Scale (RASS) ≤-2 indicates resedation
Precipitation | Initiation of remimazolam administration ~ 10 minutes after start of remimazolam
  Visually determine whether remimazolam administration causes precipitation in the fluid line through which the agent is administered
Injection pain caused by remimazolam administration | Initiation of remimazolam administration ~ 3 minutes after start of remimazolam
  Question the patient to determine if pain occurs at the intravenous site where remimazolam is administered (check only if it occurs)
Adverse events up to 48 hours after surgery | Initiation of remimazolam administration ~ 48 hours after surgery
  All adverse events including nausea/vomiting, hypertension/hypotension(30% or more change in preoperative blood pressure), bradycardia (heart rate <50 beats per minute[bpm]), tachycardia (heart rate >100 bpm)
Endogenous metabolites that occur as remimazolam is metabolized in the body (This is an exploratory check, meaning we do not know in advance what substances will be found) | Immediately before the start of remimazolam ~ 120 minutes after remimazolam cessation
  Analyze collected blood and urine to determine the metabolites of remimazolam (Therefore, various laboratory methods can be used to detect endogenous metabolites, but it is not known in advance exactly how)
Total dose of remimazolam during general anesthesia | Initiation of remimazolam administration ~ Cessation of remimazolam(up to 10 hours after start of remimazolam administration)
  Determine the total dose of remimazolam during general anesthesia
Total dose of remifentanil during general anesthesia | Initiation of remifentanil administration ~ Cessation of remifentanil(up to 10 hours after start of remifentanil administration)
  Determine the total dose of remifentanil during general anesthesia
Operation time | Start of surgery ~ End of surgery(up to 10 hours after start of surgery)
  Determine how long the surgery was performed
Anesthesia time | Initiation of remimazolam administration ~ Exit to the PACU (within 30 minutes after remimazolam cessation)
  Determine how long the general anesthesia was performed
Flumazenil dosage | Cessation of remimazolam ~ 30 minutes after remimazolam cessation
  If the participants are not awake within 10 minutes after discontinuation of remimazolam, administer flumazenil and verify the total dosage (max: 1 mg).
Pain score in PACU | PACU admission ~ PACU discharge (within 3 hours after PACU admission)
  If the participants are able to verbalize their pain, use a Numerical Rating Scale (NRS), otherwise use a Visual Analog Scale (VAS). Both scales are used to measure pain intensity on a scale of 0 to 10, with 0 being no pain and 10 being the worst pain imaginable.
Analgesic usage in PACU | PACU admission ~ PACU discharge (within 3 hours after PACU admission)
  Identify the type and dose of opioid or non-opioid pain medication used to control the participants' pain.
Delirium | After surgery ~ Hospital discharge (within 1 month after surgery)
  Determine delirium during post-operative hospitalization through electronic medical records
Postoperative complications | After surgery ~ Hospital discharge (within 1 month after surgery)
  Identify any complications during post-operative hospitalization through electronic medical records
Hospital stay after surgery | The day of surgery ~ Hospital discharge (within 1 month after surgery)
  Identify the hospital length of stay after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Byung Gun Lim, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No